CLINICAL TRIAL: NCT04208152
Title: A First-in-Human Study to Assess the Safety, Tolerability and Pharmacokinetics of anle138b in Healthy Male and Female Subjects
Brief Title: A First-in-Human Study of Single and Multiple Doses of anle138b in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MODAG GmbH (Industry)
Collaborators: Quotient Sciences (Industry); Aptuit (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: anle138b-P1-01; 2019-004218-33 (EudraCT Number)
Record Dates: First submitted 2019-12-16; First posted 2019-12-23 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: Healthy Volunteers
Keywords: anle138b; alpha-Synuclein; Oligomer modulator; Parkinson Disease; Multiple System Atrophy; Neurodegenerative diseases; Alzheimer Disease; Tauopathies; Amyloid
MeSH Terms: conditions — Parkinson Disease 4, Autosomal Dominant Lewy Body; Parkinson Disease; Multiple System Atrophy; Neurodegenerative Diseases; Alzheimer Disease; Tauopathies | interventions — 3-(1,3-benzodioxol-5-yl)-5-(3-bromophenyl)-1H-pyrazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study is double-blind. Treatment assignment will not be known to the subjects, the sponsor or the staff who are involved in the clinical evaluation of the subjects and the analysis of data. The randomisation schedule and disclosure envelopes will be generated by an unblinded statistician at Quotient Sciences.
  The FES is an open label study which includes a randomized sequence of fasted and fed state.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- anle138b (Active Comparator): Dosage: 50 mg and higher Dosage form: capsule Frequency: once daily Duration: One day for SAD and seven days for MAD
  Interventions: Drug: anle138b
- placebo (Placebo Comparator): Matching placebo Dosage form: capsule Frequency: once daily Duration: One day for SAD and seven days for MAD
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: anle138b — capsule containing excipient and anle138b
  Arms: anle138b
Drug: Placebo — matching placebo capsule containing excipient
  Arms: placebo

SUMMARY:
The purpose of this study is to determine the safety, tolerability and blood levels of orally administered anle138b in healthy subjects.

DETAILED DESCRIPTION:
This is a single-centre, study of double-blind, randomised, placebo-controlled single ascending doses (SAD) and multiple ascending doses (MAD) of anle138b in healthy subjects in study Parts 1 and 2. In study Part 3 the effect of food (FES) on the safety and PK of anle138b in healthy subjects is examined.

In the SAD cohorts, subjects will be randomly assigned to receive a single oral dose of active investigational medicinal product (IMP) or matching placebo in a sequential escalating manner with sufficient time planned between dose groups to allow interim review of the data.

In the MAD cohorts, subjects will be randomly assigned to receive oral doses of active IMP or matching placebo once daily (QD) for 7 days, in a sequential escalating manner with sufficient time planned between dose groups to allow interim review of the data.

In the FES, the effect of food on the safety and PK of anle138b is explored by administering a single dose of IMP after a high-fat breakfast. Subjects will be randomly assigned to one of 2 treatment sequence to receive anle138b in the fed or fasted state over 2 periods.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males or women of no child bearing potential
2. Age 18 to 55 years of age at the time of signing informed consent
3. Body mass index (BMI) of 18.5 to 30.0 kg/m2 as measured at screening
4. Must be willing and able to communicate and participate in the whole study
5. Must provide written informed consent
6. Must agree to adhere to the contraception requirements defined in Section 9.4
7. In the investigator's opinion, subject is able to understand the nature of the study and any risks involved in participation, and willing to cooperate and comply with the protocol restrictions and requirements.

Exclusion Criteria:

1. Subjects who have received any IMP in a clinical research study within the 90 days prior to Day 1.
2. Subjects who are study site employees, or immediate family members of a study site or sponsor employee.
3. Subjects who have previously been enrolled in this study. Subjects who have taken part in Part 1 are not permitted to take part in Part 2 or Part 3; subjects who have taken part in Part 2 are not permitted to take part in Part 3.
4. History of any drug or alcohol abuse in the past 2 years.
5. Regular alcohol consumption in males >21 units per week and females >14 units per week (1 unit = ½ pint beer, or a 25 mL shot of 40% spirit, 1.5 to 2 units = 125 mL glass of wine, depending on type).
6. A confirmed positive alcohol breath test at screening or admission.
7. Current smokers and those who have smoked within the last 12 months. A confirmed breath carbon monoxide reading of greater than 10 ppm at screening or admission.
8. Current users of e-cigarettes and nicotine replacement products and those who have used these products within the last 12 months.
9. Females of childbearing potential including those who are pregnant or lactating (all female subjects must have a negative urine pregnancy test at screening and serum pregnancy test on admission). A woman is considered of childbearing potential unless she is permanently sterile (hysterectomy, bilateral salpingectomy and bilateral oophorectomy) or is postmenopausal (had no menses for 12 months without an alternative medical cause and a serum follicle stimulating hormone concentration ≥40 IU/L).
10. Subjects with pregnant or lactating partners.
11. Subjects who do not have suitable veins for multiple venepunctures/cannulation as assessed by the investigator or delegate at screening.
12. Clinically significant abnormal clinical chemistry, haematology or urinalysis as judged by the investigator (laboratory parameters are listed in Appendix 1). Subjects with Gilbert's Syndrome are allowed. In addition the ALT and gamma glutamyl transferase (GGT) concentrations should not exceed the upper limit of normal (ULN) at screening and admission.
13. Confirmed positive drugs of abuse test result (drugs of abuse tests are listed in Appendix 1) at screening or admission.
14. Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) results
15. Evidence of renal impairment at screening, as indicated by an estimated creatinine clearance of <70 mL/min using the Cockcroft-Gault equation.
16. History of clinically significant cardiovascular, renal, hepatic, chronic respiratory or gastrointestinal disease, neurological or psychiatric disorder, as judged by the investigator.
17. Serious adverse reaction or serious hypersensitivity to any drug or the IMP excipients.
18. Presence or history of clinically significant allergy requiring treatment, as judged by the investigator. Hay fever is allowed unless it is active.
19. Donation or loss of greater than 400 mL of blood within the previous 3 months.
20. Subjects who are taking, or have taken, any prescribed or over-the-counter drug or herbal remedies (other than 4 g of paracetamol per day or HRT) in the 14 days before IMP administration (See Section 11.4). Exceptions may apply on a case by case basis, if considered not to interfere with the objectives of the study, as determined by the PI.
21. Failure to satisfy the investigator of fitness to participate for any other reason.
22. In Part 3, subjects must be able to eat 90% of the US Food and Drug Administration (FDA)-approved high-fat breakfast, including bacon.
23. Subjects with a previous history of difficulty in swallowing tablets or capsules, or an anticipated problem with swallowing a large number of capsules.
24. Blood pressure (supine) at Screening or admission outside the range: 90 to 140 mmHg for subjects <45 years or 90 to 160 mmHg for subjects >45 years for systolic BP or 40 to 90 mmHg for diastolic BP; and pulse rate outside the range of 40 to 100 bpm, unless deemed not clinically significant by the investigator and the sponsor's medical monitor.
25. Subjects with a history of cholecystectomy or gall stones.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2019-12-06 (Actual); Primary Completion 2020-08-04 (Actual); Study Completion 2020-08-04 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events in healthy volunteers with single ascending doses of anle138b (Part 1) | Day 1 to day 30 post dose
  Adverse events (AEs)
Incidence of treatment-emergent changes in clinical laboratory parameters in healthy volunteers with single ascending doses of anle138b (Part 1) | Day 1 to day 7 post dose
  clinical laboratory tests including hematology and clinical chemistry including renal function tests, hepatic enzymes, electrolytes and creatine kinase
Incidence of treatment-emergent changes in vital signs in healthy volunteers with single ascending doses of anle138b (Part 1) | Day 1 to day 7 post dose
  Blood pressure, heart rate, oral temperature
Incidence of treatment-emergent ECG changes in healthy volunteers with single ascending doses of anle138b (Part 1) | Day 1 to day 7 post dose
  Electrocardiogram (ECG) parameters including QT interval corrected for heart rate using Fridericia's formula (QTcF)
Incidence of treatment-emergent changes in physical examination in healthy volunteers with single ascending doses of anle138b (Part 1) | Day 1 to day 7 post dose
  physical examination findings
Incidence of treatment-emergent adverse events in healthy volunteers with multiple ascending doses of anle138b (Part 2) | Day 1 to day 30 post dose
  Adverse events (AEs)
Incidence of treatment-emergent changes in clinical laboratory parameters in healthy volunteers with multiple ascending doses of anle138b (Part 2) | Day 1 to day 7 post dose
  clinical laboratory tests including hematology and clinical chemistry including renal function tests, hepatic enzymes, electrolytes and creatine kinase
Incidence of treatment-emergent changes in vital signs in healthy volunteers with multiple ascending doses of anle138b (Part 2) | Day 1 to day 7 post dose
  Blood pressure, heart rate, oral temperature
Incidence of treatment-emergent ECG changes in healthy volunteers with multiple ascending doses of anle138b (Part 2) | Day 1 to day 7 post dose
  Electrocardiogram (ECG) parameters including QT interval corrected for heart rate using Fridericia's formula (QTcF)
Incidence of treatment-emergent changes in physical examination in healthy volunteers with multiple ascending doses of anle138b (Part 2) | Day 1 to day 7 post dose
  physical examination findings
Incidence of treatment-emergent adverse events in healthy volunteers with a single dose of anle138b both the fasted and fed state (Part 3) | Day 1 to day 30 post dose.
  Adverse events (AEs)
Incidence of treatment-emergent changes in clinical laboratory parameters in healthy volunteers with a single dose of anle138b both in the fasted and in the fed state (Part 3) | Day 1 to day 7 post dose
  clinical laboratory tests including hematology and clinical chemistry including renal function tests, hepatic enzymes, electrolytes and creatine kinase
Incidence of treatment-emergent changes in vital signs in healthy volunteers with a single dose of anle138b both in the fasted and in the fed state (Part 3) | Day 1 to day 7 post dose
  Blood pressure, heart rate, oral temperature
Incidence of treatment-emergent ECG changes in healthy volunteers with a single dose of anle138b both in the fasted and in the fed state (Part 3) | Day 1 to day 7 post dose
  Electrocardiogram (ECG) parameters including QT interval corrected for heart rate using Fridericia's formula (QTcF)
Incidence of treatment-emergent changes in physical examination in healthy volunteers with single ascending doses of anle138b both in the fasted and in the fed state (Part 3) | Day 1 to day 7 post dose
  physical examination findings

SECONDARY OUTCOMES:
Oral pharmacokinetics (PK) of single (Part 1) ascending doses of anle138b in the fasted state | From dosing to 48 hours post dosing
  Time prior to the first measurable concentration of anle138b.
  Time prior to the first measurable concentration of anle138b.
Oral pharmacokinetics (PK) of single (Part 1) ascending doses of anle138b in the fasted state | From dosing to 48 hours post dosing
  Time of maximum observed concentration of anle138b.
Oral pharmacokinetics (PK) of single (Part 1) ascending doses of anle138b in the fasted state | From dosing to 48 hours post dosing
  Maximum observed concentration of anle138b.
Oral pharmacokinetics (PK) of single (Part 1) ascending doses of anle138b in the fasted state | From dosing to 48 hours post dosing
  Area under the curve from 0 time to 24 h post-dose of anle138b.
Oral pharmacokinetics (PK) of single (Part 1) ascending doses of anle138b in the fasted state | From dosing to 48 hours post dosing
  Area under the curve from 0 time to the last measurable concentration of anle138b.
Oral pharmacokinetics (PK) of single (Part 1) ascending doses of anle138b in the fasted state | From dosing to 48 hours post dosing
  Area under the curve from 0 time extrapolated to infinity of anle138b levels.
Oral pharmacokinetics (PK) of single (Part 1) ascending doses of anle138b in the fasted state | From dosing to 48 hours post dosing
  Percentage of area under the curve (0-inf) extrapolated beyond the last measurable concentration of anle138b.
Oral pharmacokinetics (PK) of single (Part 1) ascending doses of anle138b in the fasted state | From dosing to 48 hours post dosing
  Slope of the apparent elimination phase of anle138b.
Oral pharmacokinetics (PK) of single (Part 1) ascending doses of anle138b in the fasted state | From dosing to 48 hours post dosing
  Apparent elimination half-life of anle138b.
Oral pharmacokinetics (PK) of single (Part 1) ascending doses of anle138b in the fasted state | From dosing to 48 hours post dosing
  Mean residence time from 0 time to the last measurable concentration after extravascular administration of anle138b.
Oral pharmacokinetics (PK) of single (Part 1) ascending doses of anle138b in the fasted state | From dosing to 48 hours post dosing
  Mean residence time extrapolated to infinity after extravascular administration of anle138b.
Oral pharmacokinetics (PK) of multiple (Part 2) ascending doses of anle138b in the fasted state | Day 1 to day 9
  Time of maximum observed concentration of anle138b
Oral pharmacokinetics (PK) of multiple (Part 2) ascending doses of anle138b in the fasted state | Day 1 to day 9
  Maximum observed concentration of anle138b
Oral pharmacokinetics (PK) of multiple (Part 2) ascending doses of anle138b in the fasted state | Day 1 to day 9
  Area under the curve over the dosing interval from time 0 to tau of anle138b
Oral pharmacokinetics (PK) of multiple (Part 2) ascending doses of anle138b in the fasted state | Day 7 to day 9
  Slope of the apparent elimination phase (last dose only) of anle138b
Oral pharmacokinetics (PK) of multiple (Part 2) ascending doses of anle138b in the fasted state | Day 1 to day 9
  Apparent elimination half-life (last dose only) of anle138b
Oral pharmacokinetics (PK) of single (Part 1) and multiple (Part 2) ascending doses of anle138b in the fasted state | Day 1 to day 9
  Accumulation Ratio based on Cmax repeated dose /Cmax single dose of anle138b
Oral pharmacokinetics (PK) of single (Part 1) and multiple (Part 2) ascending doses of anle138b in the fasted state | Day 1 to day 9
  Accumulation Ratio based on area under the curve (0 tau) repeated dose/AUC(0 tau) single dose of anle138b
Oral pharmacokinetics (PK) (Part 3) for anle138b in the fed and fasted states. | From dosing to 48 hours post dosing
  Maximum observed concentration of anle138b.
Oral pharmacokinetics (PK) (Part 3) for anle138b in the fed and fasted states. | From dosing to 48 hours post dosing
  Area under the curve from 0 time to the last measurable concentration of anle138b.
Oral pharmacokinetics (PK) (Part 3) for anle138b in the fed and fasted states | From dosing to 48 hours post dosing
  Area under the curve from 0 time extrapolated to infinity of anle138b levels.
Oral pharmacokinetics (PK) (Part 3) for anle138b in the fed and fasted states | From dosing to 48 hours post dosing
  Percentage of area under the curve (0-inf) extrapolated beyond the last measurable concentration of anle138b.

CONTACTS AND LOCATIONS:
Overall Officials: Nand Singh, BSc, MD, DPM, MFPM, Principal Investigator — Quotient Sciences Mere Way Ruddington Fields Ruddington Nottingham NG11 6JS, UK
Locations (1):
- Quotient Sciences, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wagner J, Ryazanov S, Leonov A, Levin J, Shi S, Schmidt F, Prix C, Pan-Montojo F, Bertsch U, Mitteregger-Kretzschmar G, Geissen M, Eiden M, Leidel F, Hirschberger T, Deeg AA, Krauth JJ, Zinth W, Tavan P, Pilger J, Zweckstetter M, Frank T, Bahr M, Weishaupt JH, Uhr M, Urlaub H, Teichmann U, Samwer M, Botzel K, Groschup M, Kretzschmar H, Griesinger C, Giese A. Anle138b: a novel oligomer modulator for disease-modifying therapy of neurodegenerative diseases such as prion and Parkinson's disease. Acta Neuropathol. 2013 Jun;125(6):795-813. doi: 10.1007/s00401-013-1114-9. Epub 2013 Apr 19. PMID 23604588
- [Background] Levin J, Schmidt F, Boehm C, Prix C, Botzel K, Ryazanov S, Leonov A, Griesinger C, Giese A. The oligomer modulator anle138b inhibits disease progression in a Parkinson mouse model even with treatment started after disease onset. Acta Neuropathol. 2014 May;127(5):779-80. doi: 10.1007/s00401-014-1265-3. Epub 2014 Mar 11. No abstract available. PMID 24615514
- [Background] Heras-Garvin A, Weckbecker D, Ryazanov S, Leonov A, Griesinger C, Giese A, Wenning GK, Stefanova N. Anle138b modulates alpha-synuclein oligomerization and prevents motor decline and neurodegeneration in a mouse model of multiple system atrophy. Mov Disord. 2019 Feb;34(2):255-263. doi: 10.1002/mds.27562. Epub 2018 Nov 19. PMID 30452793
- [Background] Wegrzynowicz M, Bar-On D, Calo' L, Anichtchik O, Iovino M, Xia J, Ryazanov S, Leonov A, Giese A, Dalley JW, Griesinger C, Ashery U, Spillantini MG. Depopulation of dense alpha-synuclein aggregates is associated with rescue of dopamine neuron dysfunction and death in a new Parkinson's disease model. Acta Neuropathol. 2019 Oct;138(4):575-595. doi: 10.1007/s00401-019-02023-x. Epub 2019 May 31. PMID 31165254
- [Background] Wagner J, Krauss S, Shi S, Ryazanov S, Steffen J, Miklitz C, Leonov A, Kleinknecht A, Goricke B, Weishaupt JH, Weckbecker D, Reiner AM, Zinth W, Levin J, Ehninger D, Remy S, Kretzschmar HA, Griesinger C, Giese A, Fuhrmann M. Reducing tau aggregates with anle138b delays disease progression in a mouse model of tauopathies. Acta Neuropathol. 2015 Nov;130(5):619-31. doi: 10.1007/s00401-015-1483-3. Epub 2015 Oct 6. PMID 26439832
- [Background] Martinez Hernandez A, Urbanke H, Gillman AL, Lee J, Ryazanov S, Agbemenyah HY, Benito E, Jain G, Kaurani L, Grigorian G, Leonov A, Rezaei-Ghaleh N, Wilken P, Arce FT, Wagner J, Fuhrmann M, Caruana M, Camilleri A, Vassallo N, Zweckstetter M, Benz R, Giese A, Schneider A, Korte M, Lal R, Griesinger C, Eichele G, Fischer A. The diphenylpyrazole compound anle138b blocks Abeta channels and rescues disease phenotypes in a mouse model for amyloid pathology. EMBO Mol Med. 2018 Jan;10(1):32-47. doi: 10.15252/emmm.201707825. PMID 29208638
- [Derived] Levin J, Sing N, Melbourne S, Morgan A, Mariner C, Spillantini MG, Wegrzynowicz M, Dalley JW, Langer S, Ryazanov S, Leonov A, Griesinger C, Schmidt F, Weckbecker D, Prager K, Matthias T, Giese A. Safety, tolerability and pharmacokinetics of the oligomer modulator anle138b with exposure levels sufficient for therapeutic efficacy in a murine Parkinson model: A randomised, double-blind, placebo-controlled phase 1a trial. EBioMedicine. 2022 Jun;80:104021. doi: 10.1016/j.ebiom.2022.104021. Epub 2022 Apr 29. PMID 35500536
- See also: MODAG GmbH - Sponsor homepage — http://www.modag.net/index.php/en/